CLINICAL TRIAL: NCT02291809
Title: REMUNE HIV/AIDS Vaccine Phase II Pediatric Safety & Efficacy Clinical Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Immune Response BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR-HIV-007
Record Dates: First submitted 2014-11-06; First posted 2014-11-14 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Pediatric; Vaccine; HIV-1 Immunogen
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — remune; HIV-1 immunogen, incomplete Freund's adjuvant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- REMUNE (Experimental): Remune vaccine consists of a suspension of killed HIV-1 virus particles that have been emulsified with Incomplete Freund's Adjuvant (IFA, a mixture of mannide mono-oleate and a highly purified mineral oil). Each dose is given by IM injection and contains 10 μg of p24 antigen in approximately 100 μg of total protein.
  Interventions: Biological: REMUNE
- REMUNE Low Dose (Placebo Comparator): Remune low dose vaccine consists of a suspension of killed HIV-1 virus particles that have been emulsified with Incomplete Freund's Adjuvant (IFA, a mixture of mannide mono-oleate and a highly purified mineral oil). Each dose is given by IM injection and contains 2.5 μg of p24 antigen in approximately 25 μg of total protein.
  Interventions: Biological: REMUNE

INTERVENTIONS:
Biological: REMUNE — Inoculation of HIV-1 Virus via Vaccination of Whole Killed GP120 Depleted P24 Antigen Vaccine
  Other Names: HIV-1 Immunogen

SUMMARY:
The primary objective is to compare & evaluate between the treatment groups the changes in decline/reduction of HIV viral load & increase changes in WBC white blood cell counts in the adult Remune dose vs the low dose Remune placebo groups. Additional objectives include changes in CD4+ & CD8+ T cell counts along with increased HIV immunity.

DETAILED DESCRIPTION:
This is a 26 subject Multi Center double-blind randomized, Safety & Efficacy, pediatric HIV/AIDS Phase II study, to primarily to evaluate the safety and efficacy of HIV-1 immunogen and secondarily to examine changes in CD4+ & CD8+ T cell counts, determine Remune vaccines effect of multiple inoculations of HIV-1 immunogen on viral replication in children with HIV-1 infection & immunogenicity of Remune. Multi-center, randomized , double-blind, placebo-controlled, two arm parallel design study of Remune.

ELIGIBILITY:
Inclusion Criteria:

* Children clinically diagnosed with HIV that are 3 months of age to the age 16 years old
* Subjects on any approved FDA antiviral medication except triple cocktail HAART drugs

Exclusion Criteria:

* Truvada
* Triple cocktail HAART drugs
* Healthy subjects

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2017-11; Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to compare & evaluate between the treatment groups the changes in HIV viral load at Week 52 | 52 Weeks
  The primary objective is to compare & evaluate between the treatment groups the changes in HIV viral load (HIV RNA Viral Load) at Week 52
The primary objective is to compare & evaluate between the treatment groups the changes in WBC white blood cell counts at Week 52 | 52 Weeks
  The primary objective is to compare & evaluate between the treatment groups the changes in WBC white blood cell counts at Week 52

SECONDARY OUTCOMES:
The secondary objective is to evaluate & compare changes in CD4+ & CD8+ T cell counts between the treatment groups | 52
  The secondary objective is to evaluate & compare changes in CD4+ & CD8+ T cell counts between the treatment groups
The secondary objective is to evaluate & compare the effect of multiple inoculations of HIV-1 immunogen on viral replication in children with HIV-1 infection | 52 Weeks
  HIV-1 immunogen on viral replication in children with HIV-1 infection
The secondary objective is to evaluate & compare between the treatment groups to induce immune responses between adult and low doses of REMUNE | 52 Weeks
  The secondary objective is to evaluate & compare between the treatment groups the ability to induce immune responses between the adult and low doses of REMUNE

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Bartholomew, PhD, Study Director — Immune Response BioPharma, Inc. Chief R&D Officer
Locations (1):
- Clinical Site TBA, San Diego, California, United States